CLINICAL TRIAL: NCT02017119
Title: Comparison Between Lactulose and Lactulose-Paraffin in Cirrhotic Patients: Impact on the Recurrence of Encephalopathy, Tolerance and Adherence to Treatment, Costs, and Quality of Life
Brief Title: Comparison Between Lactulose and Lactulose-Paraffin in Cirrhotic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, ALDO TORRE DELGADILLO, Principal Investigator., Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GAS-282-10/11-1
Record Dates: First submitted 2013-12-16; First posted 2013-12-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactulose (Experimental): Lactulose 15ml oral intake 8hrs daily for 6 months. The dose may be modified depending on the number of total bowel movements, (the expected range is 2 - 4 per day).
  Interventions: Drug: Comparison between Lactulose and Lactulose-Paraffin
- Lactulose-paraffin (Experimental): Paraffin 15g daily for 6 months. The dose may be modified depending on the number of total bowel movements, (the expected range is 2 - 4 per day).
  Interventions: Drug: Comparison between Lactulose and Lactulose-Paraffin

INTERVENTIONS:
Drug: Comparison between Lactulose and Lactulose-Paraffin

SUMMARY:
Hepatic encephalopathy (HE) is an important complication of liver cirrhosis. Lactulose is a first line treatment for HE, but the adherence to this treatment is relatively low, due to side effects such as diarrhea, distention, etc.

DETAILED DESCRIPTION:
Lactulose is a first line treatment for HE, but the adherence to this treatment is relatively low due to side effects. Lactulose-paraffin recently available in the market can be used for the treatment of HE, and possibly have fewer side effects.

The aim of this study was to compare the adherence of the treatment of lactulose and lactulose-paraffin.

ELIGIBILITY:
Inclusion Criteria:

* Liver cirrhosis
* History of an event of hepatic encephalopathy.
* Ambulatory patients

Exclusion Criteria:

* Alcoholism with active ingest of alcohol in the last 6 months
* Labour turn-overs
* Pregnancy
* Personal history of surgery in the last 4 weeks
* Spontaneous bacterial Peritonitis
* Use of neuropsychiatric drugs
* Neuropsychiatric disorders (Schizophrenia, bipolar disorder, major depression, dementia and Attention-deficit hyperactivity disorder)
* Thyroid disorders without replacement therapy
* Renal failure
* Hepatic or renal transplant
* Personal history of hepatocellular carcinoma
* Placement of transjugular intrahepatic portosystemic shunt
* Use of a probiotic in the last 6 month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | 6 months
  Provide evidence of better adherence to treatment with lactulose-paraffin in cirrhotic patients with a history of hepatic encephalopathy, which should be reflected in fewer hospitalizations, lower costs and better quality life.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico